CLINICAL TRIAL: NCT06445608
Title: PICANTE: PIvotal Trial of the KARDION Cory P4 MechANical Circulatory SupporT SystEm
Brief Title: PIvotal Trial of the KARDION Cory P4 MechANical Circulatory SupporT SystEm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kardion Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000001057
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease
Keywords: High-risk PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- KARDION Cory P4 System (Experimental)
  Interventions: Device: Percutaneous Mechanical Circulatory Support
- Commercial Control (Active Comparator)
  Interventions: Device: Percutaneous Mechanical Circulatory Support

INTERVENTIONS:
Device: Percutaneous Mechanical Circulatory Support — Patients are randomized to receive one of two types of percutaneous mechanical circulatory support devices during a high-risk PCI procedure.

SUMMARY:
This purpose of this trial is to demonstrate 30 day safety and effectiveness outcomes of the KARDION CORY P4 System in subjects who require hemodynamic support during a high-risk PCI procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18 and ≤ 90 years at the time of screening
2. The subject has an LV ejection fraction of < 50% (within 90 days of index procedure) AND is at high-risk due to any of the following:

   * Unprotected left main coronary artery stenosis disease
   * Last remaining epicardial native coronary artery
   * Significant three vessel coronary artery disease
   * Significant two vessel coronary artery disease of complex lesions
   * Significant single vessel coronary artery disease of complex lesions and non-treated CTO
   * Target vessel is a CTO with planned retrograde approach
   * Intended calcium modification (by atherectomy, lithotripsy or laser)

     * In multiple vessels OR
     * In the left main OR
     * In a final patent conduit OR
     * Where the anatomic SYNTAX score is ≥32
3. Local heart team (interventional cardiologist, cardiac surgeon) has determined that the subject is an appropriate candidate for a PCI supported with a Mechanical Circulatory Support (MCS) System
4. Confirmed access site vasculature greater than 5.5 mm as measured by CT or femoral duplex ultrasound
5. The subject is willing and able to comply with the protocol-specified treatment and follow-up evaluations
6. The subject has been informed of the nature of the trial, agrees to its provisions, and has provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Exclusion Criteria:

1. Any prior coronary revascularization or revascularization attempt within 30 days prior to index procedure
2. STEMI within 7 days prior to index procedure - defined as new ST elevation at the J point in at least 2 contiguous leads of ≥ 2 mm (0.2 mV) in men or ≥ 1.5 mm (0.15 mV) in women in leads V2-V3 and/or of ≥ 1 mm (0.1 mV) in other contiguous chest leads or the limb leads
3. Non-STEMI within 7 days prior to index procedure with an elevated cardiac biomarker (CK-MB or Troponin >1x ULN) without CK-MB or Troponin value down trending
4. Cardiac arrest within 7 days prior to index procedure requiring CPR or defibrillation
5. Subjects with sustained ventricular tachycardia or repetitive/ prolonged non-sustained ventricular tachycardia or complex ventricular ectopy
6. Current left ventricular thrombus
7. Significant right heart failure (right ventricular fractional area change <35% on echocardiography)
8. Known severe pulmonary hypertension (right ventricular systolic pressure (RVSP) on echo or pulmonary artery systolic pressure (PASP) on right heart catheterization > 70mmHg
9. Combined cardiorespiratory failure
10. Presence of an atrial or ventricular septal defect (including post-infarct VSD)
11. Hypertrophic obstructive cardiomyopathy (HOCM), restrictive cardiomyopathy, or constrictive pericarditis
12. Cardiogenic shock (Cardiac index < 1.8 L/min/m2)
13. Use of inotropic or pressor therapy within 72 hours of the planned index procedure. NOTE: Use of inotropic or pressor therapy for the sole purpose of blood pressure support associated with anesthesia for the procedure is acceptable.
14. Any use of mechanical circulatory support or an extracorporeal membrane oxygenation device within 14 days prior to index procedure
15. Severe aortic valve insufficiency or stenosis or aortic valve replacement
16. Clinically-relevant vascular disease that precludes the placement of a MCS device
17. Cerebrovascular Accident (CVA) within 180 days prior to index procedure
18. Transient Ischemic Attack (TIA) within 90 days prior to index procedure
19. Known or suspected coagulopathy or abnormal coagulation parameters (defined as platelet count ≤ 100,000 or spontaneous INR ≥ 1.5 or known fibrinogen ≤ 1.5 g/L)
20. Known hemoglobin diseases, such as sickle cell anemia, hemolytic anemia or thalassemia
21. Subject has evidence of an active infection on the day of the index procedure requiring oral or intravenous antibiotics
22. Active infection of the intended access site
23. Chronic renal dysfunction (eGFR < 30 mL/min/1.73 m²) and/or patients requiring renal replacement therapy with dialysis
24. KnownHistory of liver dysfunction with elevation of liver enzymes and bilirubin 3 times the upper limit of normal (ULN) within 90 days prior to index procedure
25. Known or suspected severe pulmonary disease (e.g., forced expiratory volume (FEV)1 < 1.0 L/s)
26. Allergy, sensitivity or intolerance to anesthesia, heparin, aspirin, adenosine diphosphate (ADP) receptor blockers, or contrast media, including known heparin-induced thrombocytopenia (HIT)
27. Any non-cardiac condition with life expectancy < 1 year
28. Subject is presently or recently intubated for the current admission (NOTE: recently intubated patients must be extubated for > 24 hours with full neurologic recovery). Procedure-related intubation is acceptable.
29. Decompensated heart failure requiring IV diuretics, vasopressors or inotropic support within 72 hours of index procedure
30. Patients with an organ transplant
31. Patients with implanted left ventricular assist device
32. Cardiac tamponade
33. Left ventricular rupture
34. Women who are lactating, pregnant, or plan to become pregnant during the course of the investigation
35. Any anatomical restriction that would preclude a MCS device from being delivered through the femoral artery to the left ventricle
36. Subject has other medical, social or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with trial procedures
37. Current participation in another investigational drug or device trial
38. Anticipated need for continued MCS support after conclusion of the PCI procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MACCE | 30 days post-procedure
  The primary effectiveness endpoint of the clinical investigation is a composite endpoint of major adverse cardiac and cerebrovascular events (MACCE) comprised of all-cause death, myocardial infarction, stroke/TIA, target lesion revascularization, vascular complications, major bleeding, and acute kidney injury.
Device-Related Safety | 30 days post-procedure
  The primary safety endpoint of the clinical investigation is a composite endpoint of device-related safety events (as adjudicated by the CEC) requiring intervention, including cardiac or vascular complication, limb ischemia, increase in aortic insufficiency, or CPR or ventricular arrhythmia requiring cardioversion.

SECONDARY OUTCOMES:
Technical Success | Index procedure
  Technical Success defined as the ability of the MCS System to be delivered, operated without device malfunction through the end of procedure, and successful retrieval.
Procedural Success | Index Procedure
  Procedural Success defined as Technical Success and the ability of the MCS System to provide hemodynamic support preventing severe hypotension and without the need for escalation of mechanical circulatory support (i.e., replacement of the MCS System with a higher output mechanical circulatory support device). Severe hypotension defined as requiring continuous infusion of inotropic/pressor medications to restore hemodynamics to mean arterial pressure greater than 60 mmHg.
Serious Device-Related Adverse Events | Index procedure through 30-day follow-up
  Safety Outcome defined as Serious Device-Related Adverse Events (defined as any Serious Adverse Event adjudicated as related to the device by the Clinical Events Committee (CEC)) through 30 days following the index procedure.
Individual MACCE components | Index procedure through 30-day follow-up
  Individual MACCE components: all-cause death, MI, stroke/TIA, target lesion revascularization, vascular complications, major bleeding, and acute kidney injury.
Death | Index procedure through 30-day follow-up
  Cardiovascular death and non-cardiovascular death.
Health Outcomes Measure: all-cause death | Index procedure through 30-day follow-up
  all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Samin Sharma, MD, Study Chair — Icahn School of Medicine at Mount Sinai; William Nicholson, MD, Study Chair — Emory University
Locations (18):
- United States (18):
  - Dignity Health - Chandler Regional Medical Center, Chandler, Arizona
  - HonorHealth Research and Innovation Institute, Scottsdale, Arizona
  - Arkansas Cardiology, P.A., Little Rock, Arkansas
  - North Suburban Medical Center, Thornton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Ascension St. Vincent's, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Ascension St. Vincent, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Mount Sinai, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - The Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Heart and Vascular Research at WellSpan Health, York, Pennsylvania
  - Ascension Saint Thomas, Nashville, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No